CLINICAL TRIAL: NCT02703714
Title: Phase II Trial of Pembrolizumab (MK-3475) With GM-CSF Induction in Advanced Biliary Cancers
Brief Title: Pembrolizumab and GM-CSF in Biliary Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robin Kate Kelley (Other)
Collaborators: American Society of Clinical Oncology (Other); Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Robin Kate Kelley, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 154524; NCI-2017-01372 (Other: NCI Clinical Trials Reporting Program (CTRP)); R03CA212877 (NIH)
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Results first posted 2022-01-12 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Biliary Cancer
Keywords: Advanced; Locally-advanced; Not eligible for resection; Prior chemotherapy treatment
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — pembrolizumab; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and GM-CSF (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Patients also receive sargramostim subcutaneous injection (SC) on days 1-14 of courses 1-2 or 2-3. Treatment repeats every 21 days for up to 2 courses for sargramostim and for up to 35 courses (24 months) for pembrolizumab in the absence of disease or unaccepted toxicity.
  Interventions: Drug: Pembrolizumab; Drug: Sargramostim

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg given intravenously (IV)
  Other Names: MK-3475; Keytruda
Drug: Sargramostim — 250 µg given subcutaneously (SC)
  Other Names: GM-CSF

SUMMARY:
This is an open label phase II trial to examine efficacy and safety of a novel combination of pembrolizumab plus induction GM-CSF in patients with advanced biliary cancers treated at University of California, San Francisco (UCSF).

This phase II study will examine the efficacy and safety of the novel combination of pembrolizumab plus induction GM-CSF in advanced biliary cancer patients with the hypotheses that the combination may increase proportion of patients with overall response compared to contemporary historical controls, with acceptable safety.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrate adequate organ function

  * Absolute neutrophil count (ANC) >= 1,000/microliter (mcL)(performed within 28 days of treatment initiation)
  * Platelets >= 60,000/mcL (>= 75,000/mcL in expansion cohort) (performed within 28 days of treatment initiation)
  * Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment) (performed within 28 days of treatment initiation)
  * Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl)) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (performed within 28 days of treatment initiation)
  * Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (performed within 28 days of treatment initiation)
  * Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) =< 5 X ULN (performed within 28 days of treatment initiation)
  * Albumin >= 2.5 mg/dL (performed within 28 days of treatment initiation)
  * International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as prothrombin time (PT) or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (performed within 28 days of treatment initiation)
  * Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (performed within 28 days of treatment initiation)
* Patients with known hepatitis B (HBV) or hepatitis C virus (HCV) infection are eligible provided liver function parameters meet laboratory eligibility criteria
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

ADDITIONAL EXPANSION COHORT SUBJECT INCLUSION CRITERIA

* Tumor measurable by RECIST 1.1 including >= 1 target lesion not planned for biopsy
* Presence of >= 1 tumor lesion not included as a RECIST 1.1 target lesion which is assessed by investigator and/or radiologist as likely to be amenable to percutaneous biopsy by punch, computed tomography (CT)-, or ultrasound-guided core needle biopsy for serial sampling on treatment
* Platelet count >= 75,000/mcL
* No contraindication to tumor biopsy at time of study enrollment
* Consent for on-treatment paired biopsies

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated and received study therapy in a study of an investigational agent, or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy for purposes of immunosuppression or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active Bacillus Tuberculosis (TB).
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has untreated active Hepatitis B (e.g., HBsAg reactive).
* Has an active infection requiring systemic antibiotic therapy at time of enrollment.

  • Treatment with antibiotic prophylaxis for indwelling biliary stent(s) or peri-procedural antibiotics for uncomplicated biliary stent exchanges is allowed and not an exclusion
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has received treatment with an anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has received treatment with chemotherapy, targeted small molecule therapy, or radiation therapy to non-liver sites within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent administered more than 2 weeks earlier.
* Has had prior chemoembolization, bland embolization, radioembolization, local ablative therapies, radiation to liver tumors, or major surgery such as liver resection within 4 weeks prior to study enrollment or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to intervention more than 4 weeks earlier.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of or any evidence of active, non-infectious pneumonitis.
* Has had prior liver or other organ transplantation.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Kate Kelley, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keenan BP, McCarthy EE, Ilano A, Yang H, Zhang L, Allaire K, Fan Z, Li T, Lee DS, Sun Y, Cheung A, Luong D, Chang H, Chen B, Marquez J, Sheldon B, Kelley RK, Ye CJ, Fong L. Circulating monocytes associated with anti-PD-1 resistance in human biliary cancer induce T cell paralysis. Cell Rep. 2022 Sep 20;40(12):111384. doi: 10.1016/j.celrep.2022.111384. PMID 36130508

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab and GM-CSF
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab and GM-CSF
Number analyzed (Participants) | 42
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 1
  40-49 years old | 3
  50-59 years old | 15
  60-69 years old | 12
  70-79 years old | 10
  80-89 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 42
Biliary Cancer Sub-types [Count of Participants; unit: Participants] — Intrahepatic bile duct cancer forms in the bile ducts inside the liver. Extrahepatic bile duct cancer forms in the bile ducts outside the liver. Gallbladder Cancer forms in the gallbladder itself.
  Participants
    Intrahepatic Cholangiocarcinoma (ICC) | 28
    Extrahepatic Cholangiocarcinoma (ECC) | 11
    Gallbladder Cancers (GBC) | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Proportion of subjects with measurable disease at study entry who obtained either a complete response (CR) or partial response (PR) (confirmed + unconfirmed) using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 at any time during the course of treatment.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Pembrolizumab and GM-CSF
Number analyzed (Participants) | 42
proportion of participants | 0.12 [0.04 to 0.26]

2. Secondary Outcome: Proportion of Participants With Treatment-related AEs
Description: Safety events will be summarized based on proportion of total subjects, by preferred term. Only treatment-related >=grade 3 Adverse Events (AE)s will be reported.
Time Frame: During study treatment and for 30 days after last dose or until start of new treatment (up to 2 years)
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Pembrolizumab and GM-CSF
Number analyzed (Participants) | 42
proportion of participants | 0.095 [0.03 to 0.23]

3. Secondary Outcome: Proportion of Participants With PD-L1 Positive Status
Description: PD-L1 expression will be measured by immunohistochemistry (IHC) and classified as positive or negative by central laboratory testing (QualTek Laboratories) using pre-specified cut-points; will be reported along with 95% confidence interval (CI)
Time Frame: Up to 4 years
Population: Only 28 participants had lab data collected for this endpoint
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Pembrolizumab and GM-CSF
Number analyzed (Participants) | 28
proportion of participants | 0.36 [0.19 to 0.56]

4. Secondary Outcome: Proportion of Participants With Progression-Free Survival (PFS) at 6 Months
Description: Proportion of participants with PFS Time from date of first dose of protocol therapy to date of first documented radiographic and/or clinical disease progression per RECIST version 1.1 or death from any cause
Time Frame: 6 months after start of study treatment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Pembrolizumab and GM-CSF
Number analyzed (Participants) | 42
proportion of participants | 0.26 [0.14 to 0.42]

5. Secondary Outcome: Median Duration of Response
Description: Time from first documented evidence of CR or PR until the first documented sign of disease progression or death
Time Frame: Within 4 years after start of study treatment
Population: Only 5 participants demonstrated an overall response
Measure: Median (Full Range); unit: days
Arm/Group | Pembrolizumab and GM-CSF
Number analyzed (Participants) | 5
days | 294 [144 to 1379]

6. Secondary Outcome: Median Duration of Response Stratified by Sub-type of Biliary Cancer
Description: Time from first documented evidence of CR or PR until the first documented sign of disease progression or death stratified by sub-type of biliary cancer
Time Frame: Within 4 years after start of study treatment
Population: Only 5 participants demonstrated a response of CR or PR, and all participants were diagnosed with Intrahepatic Cholangiocarcinoma (ICC)
Measure: Median (Full Range); unit: days
Arm/Group | Pembrolizumab and GM-CSF
Number analyzed (Participants) | 5
days
  Intrahepatic Cholangiocarcinoma (ICC) | 294 [144 to 1379]
  Extrahepatic Cholangiocarcinoma (ECC): number analyzed (Participants) | 0
  Gallbladder Cancer (GBC): number analyzed (Participants) | 0

7. Secondary Outcome: Median Progression Free-Survival (PFS)
Description: Time from date of first dose of protocol therapy to date of first documented radiographic and/or clinical disease progression per RECIST version 1.1 or death from any cause
Time Frame: Within 4 years after start of study treatment
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pembrolizumab and GM-CSF
Number analyzed (Participants) | 42
days | 63 [55 to 125]

8. Secondary Outcome: Median PFS Stratified by Sub-type of Biliary Cancer
Description: Time from date of first dose of protocol therapy to date of first documented radiographic and/or clinical disease progression per RECIST version 1.1 or death from any cause stratified by sub-type of biliary cancer
Time Frame: Within 4 years after start of study treatment
Population: Results are reported by sub-type of biliary cancer
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pembrolizumab and GM-CSF
Number analyzed (Participants) | 42
days
  Intrahepatic Cholangiocarcinoma (ICC): number analyzed (Participants) | 28
  Intrahepatic Cholangiocarcinoma (ICC) | 63 [53 to 175]
  Extrahepatic Cholangiocarcinoma (ECC): number analyzed (Participants) | 11
  Extrahepatic Cholangiocarcinoma (ECC) | 58 [53 to 151]
  Gallbladder Cancer (GBC): number analyzed (Participants) | 3
  Gallbladder Cancer (GBC) | 121 [57 to 132]

9. Secondary Outcome: Median Overall Survival (OS)
Description: Time from first dose of protocol therapy to the date of death due to any cause
Time Frame: Within 4 years after start of treatment
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pembrolizumab and GM-CSF
Number analyzed (Participants) | 42
days | 393 [243 to 573]

10. Secondary Outcome: Median Overall Survival (OS) Stratified by Sub-type of Biliary Cancer
Description: Time from first dose of protocol therapy to the date of death due to any cause stratified by sub-type of biliary cancer.
Time Frame: Within 4 years after start of treatment
Population: Results are reported by sub-type of biliary cancer
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pembrolizumab and GM-CSF
Number analyzed (Participants) | 42
days
  Intrahepatic Cholangiocarcinoma (ICC): number analyzed (Participants) | 28
  Intrahepatic Cholangiocarcinoma (ICC) | 424 [295 to 1033]
  Extrahepatic Cholangiocarcinoma (ECC): number analyzed (Participants) | 11
  Extrahepatic Cholangiocarcinoma (ECC) | 286 [108 to 623]
  Gallbladder Cancers (GBC): number analyzed (Participants) | 3
  Gallbladder Cancers (GBC) | 165 [156 to 393]

ADVERSE EVENTS:
Time Frame: Up to 4 years
Arm/Group | Pembrolizumab and GM-CSF
All-Cause Mortality (participants affected / at risk) | 37/42
Serious Adverse Events (participants affected / at risk) | 18/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and GM-CSF (N=42)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Biliary tract infection (Infections and infestations) | 4 (8)
Fever (General disorders) | 4 (5)
Sepsis (Infections and infestations) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (2)
Delirium (Psychiatric disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Lung Infection (Infections and infestations) | 2 (2)
Hepatic Hemorrhage (Hepatobiliary disorders) | 1 (1)
Ascities (Gastrointestinal disorders) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Extraocular muscle paresis (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and GM-CSF (N=42)
Diarrhea (Gastrointestinal disorders) | 18 (23)
Abdominal pain (Gastrointestinal disorders) | 17 (28)
Nausea (Gastrointestinal disorders) | 12 (17)
Ascites (Gastrointestinal disorders) | 11 (15)
Constipation (Gastrointestinal disorders) | 9 (9)
Vomiting (Gastrointestinal disorders) | 8 (9)
Abdominal distension (Gastrointestinal disorders) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 5 (6)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 5 (7)
Bloating (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Flatulence (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 19 (29)
Fever (General disorders) | 14 (28)
Injection site reaction (General disorders) | 14 (16)
Chills (General disorders) | 12 (13)
Edema limbs (General disorders) | 9 (11)
General disorders and administration site conditions - Other (General disorders) | 5 (5)
Non-cardiac chest pain (General disorders) | 5 (5)
Leukocytosis (Blood and lymphatic system disorders) | 30 (47)
Anemia (Blood and lymphatic system disorders) | 4 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (22)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (8)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 (25)
Anorexia (Metabolism and nutrition disorders) | 10 (12)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (17)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 (20)
Weight loss (Investigations) | 11 (14)
Aspartate aminotransferase increased (Investigations) | 7 (14)
Blood bilirubin increased (Investigations) | 6 (9)
Creatinine increased (Investigations) | 6 (6)
Platelet count decreased (Investigations) | 6 (10)
Alanine aminotransferase increased (Investigations) | 4 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (18)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Upper respiratory infection (Infections and infestations) | 10 (16)
Urinary tract infection (Infections and infestations) | 4 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (9)
Dizziness (Infections and infestations) | 4 (4)
Hypothyroidism (Endocrine disorders) | 8 (10)
Hyperthyroidism (Endocrine disorders) | 4 (5)
Palpitations (Cardiac disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Dry eye (Eye disorders) | 5 (6)
Depression (Psychiatric disorders) | 3 (4)
Confusion (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT02703714/Prot_SAP_000.pdf